CLINICAL TRIAL: NCT06956274
Title: Ostomy Readmission Reduction Program
Status: Not yet recruiting | Type: Observational
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Yosef Nasseri, MD, Colon and Rectal Surgeon, Cedars-Sinai Medical Center
Other Study IDs: STUDY00003920
Record Dates: First submitted 2025-04-16; First posted 2025-05-04 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-04

CONDITIONS: Ostomy - Ileostomy or Colostomy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Preoperative Telehealth — Conduct a preoperative telehealth consultation with a Certified Wound, Ostomy, and Continence Nurse (WOCN) to provide patient education on post-surgical care expectations.
Other: Measure Ostomy Output — Patients will be sent home with a measuring container (graduated container) and will measure their ostomy output every 12 hours and record it in a pad that will be provided to them.

SUMMARY:
The purpose of this study is to reduce complications like peristomal skin issues, stoma-related problems, dehydration, and other preventable factors that can lead to re-hospitalization within the first 30 days after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Elective operations involving an ileostomy or a colostomy
* Individuals 18 years old or older are included

Exclusion Criteria:

* Individuals under age 18
* Pregnant patients
* Emergency operations
* Patients with existing pre operative ostomies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will be identified from our outpatient clinic during surgical consultations.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Readmission to hospital within 30 Days of Surgery | 30 Days Post Surgery
  The proportion of participants who are readmitted to the hospital within 30 days following surgery. Readmissions will be evaluated for any reason, including complications, adverse events, or recovery issues that necessitate hospitalization after the initial surgical procedure.

SECONDARY OUTCOMES:
Hospital Length of Stay | From index surgery to discharge (up to 30 days postoperatively)
  Total duration of hospitalization from the time of the index surgery until discharge.
Incidence of Acute Kidney Injury (AKI) | From index surgery through 30 days postoperatively
  Number of participants who develop AKI, defined as an increase in serum creatinine of ≥0.3 mg/dL from baseline, during index admission or upon 30-day readmission.
Incidence of Peristomal Skin Complications | From index surgery through 30 days postoperatively
  Number of participants who develop peristomal skin problems (e.g., irritation, excoriation, or dermatitis) during the index admission or within 30 days postoperatively.
Incidence of Stoma-Related Leakage | From index surgery through 30 days postoperatively
  Number of participants who experience unintended escape of stoma output (leakage) during index admission or within 30 days postoperatively.

CONTACTS AND LOCATIONS:
Overall Officials: Yosef Nasseri, MD, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Surgery Group LA, Los Angeles, California, United States